CLINICAL TRIAL: NCT06231862
Title: Gene Expression Objective Definition of Early Sepsis In Children
Acronym: GEODESIC
Status: Completed | Type: Observational
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Immunexpress (Industry)
Responsible Party: Sponsor
Other Study IDs: STUDY00001733
Record Dates: First submitted 2024-01-21; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Sepsis; Non-Infectious Systemic Inflammatory Response Syndrome
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Paired blood samples for paired mRNA expression analysis, the first around the time of PICU admission and the second around 48 hours later

GROUPS / COHORTS (3):
- Suspected/documented bacterial sepsis: Patients have evidence of an acute bacterial infection with organ dysfunction
  Interventions: Diagnostic Test: SeptiCyte (various)
- Suspected/documented viral sepsis: Patients have evidence of an acute viral infection with organ dysfunction
  Interventions: Diagnostic Test: SeptiCyte (various)
- Infection negative systemic inflammation (SIRS): Patients have no active infection but exhibit SIRS
  Interventions: Diagnostic Test: SeptiCyte (various)

INTERVENTIONS:
Diagnostic Test: SeptiCyte (various) — mRNA expression scores

SUMMARY:
GEODESIC is a prospective descriptive cohort investigation that will examine the generalizability of the novel host gene expression biomarkers, SeptiCyteTM LAB, SeptiCyteTM VIRUS, SeptiCyteTM BACT, and SeptiCyteTM TRIAGE (collectively 18 genes or SeptiCyteTM LVBT) and SeptiCyteTM RAPID, for differentiating children with bacterial sepsis, versus severe viral illness, versus non-infectious related systemic inflammatory response syndrome.

DETAILED DESCRIPTION:
Specific Aim 1. Validate the robustness of the SeptiCyteTM LVBT gene expression signatures for providing clear discrimination between critically ill children with bacterial sepsis versus severe viral illness versus infection-negative systemic inflammation (INSI) secondary to a variety of etiologies.

Approach: We will expand our previous Genotypes And Phenotypes in Pediatric SIRS and Sepsis (GAPPSS) INSI cohort to children with recent trauma, thermal burns, anoxic-ischemic reperfusion events, exposure to cardiopulmonary bypass, extracorporeal life support, or dialytic therapy, CAR-T cell therapy, and various rheumatologic diagnoses. e we will recruit children with bacterial and viral infection who demonstrate a spectrum of illness severity and organ dysfunction. This specific aim will demonstrate the generalizability of SeptiCyteTM LVBT among critically children with life-threatening infectious disease or INSI.

Specific Aim 2. Determine if SeptiCyteTM LVBT gene expression signatures trend towards resolution of previously induced or suppressed gene expression states as critical illness resolves.

Approach: We will obtain paired blood samples for SeptiCyteTM LVBT gene expression, the first around the time of intensive care unit (ICU) admission (critically ill) and the second at ICU discharge approximately 48 hours later (transition to acute care). Resolution of critical illness will be quantified by serial daily measures of composite organ dysfunction.

Specific Aim 3. Ascertain that performance of SeptiCyteTM RAPID utilizing a point of care device at Seattle Children's will be equivalent to centralized assessment using SeptiCyteTM LAB.

Approach: Blood samples will be processed on site (Seattle Children's) for SeptiCyte RAPID testing. SeptiCyteTM RAPID is the result of the translation of the SeptiCyteTM LAB test to the cartridge-based Biocartis Idylla™ platform.

ELIGIBILITY:
Inclusion Criteria:

INSI Cohort

* Admitted to the PICU
* New severe trauma OR
* New thermal burns OR
* Rheumatologic diagnoses OR
* Post-initiation (or circuit change) of extracorporeal life support OR
* Post anoxic-ischemic-reperfusion insults OR
* Infants undergoing cardiac surgery with cardiopulmonary bypass OR
* CAR-T cell therapy
* Parents speak English or Spanish AND
* Not previously enrolled in the GEODESIC investigation

Pediatric Bacterial Sepsis Cohort

* Admitted to the PICU
* Parents speak English or Spanish AND
* Exhibit SIRS criteria including at least fever/hypothermia or leukocytosis/leukopenia or left shift on the leukocyte differential AND
* Strongly suspected or documented source of bacterial infection per primary care team
* Not previously enrolled in the GEODESIC investigation

Pediatric Bacterial Sepsis Cohort

* Admitted to the PICU
* Parents speak English or Spanish AND
* Positive PCR or culture verifying a viral infection
* Not previously enrolled in the GEODESIC investigation

Exclusion Criteria:

* Not expected to survive the PICU stay
* Child has 'ward of the state' status

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Critically ill children with systemic inflammatory response secondary to bacterial or viral sepsis or non-infectious SIRS
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
mRNA expression | At PICU admission and 48 hours later
  SeptiCyte (various) gene expression scores

CONTACTS AND LOCATIONS:
Overall Officials: Jerry J Zimmerman, MD, PhD, Principal Investigator — Seattle Children's Research Center
Locations (2):
- United States (2):
  - Seattle Children's Hospital, Harborview Medical Center, Seattle, Washington
  - Seattle Children's Hospital, Seattle, Washington